# Exploring Merkel Cell Carcinoma Clinical Trial Engagement Patterns: Unveiling Participation Trends Among Individuals Affected by the Condition

An Informed Consent Form For Patients With Merkel Cell Carcinoma in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: September 8, 2023

Introduction to the Informed Consent Document

If you are given the task of completing this form, it suggests your prospective inclusion in an observational clinical trial intended exclusively for those dealing with Merkel cell carcinoma. This paper is a detailed handbook that reveals the study's main aims, thorough implementation strategy, and numerous ramifications, both good and potentially negative. Before making a choice, it is critical to think about your prospective involvement carefully, and obtaining advice from a trustworthy confidant can provide vital insights. If any of the material presented here is confusing, or if you have any questions, please know that the researcher is accessible to answer them.

# Study Aim

Merkel cell carcinoma (MCC) is a rare and aggressive type of skin cancer. It develops from Merkel cells, which are specialized cells located in the top layer of the skin (the epidermis). These cells are responsible for the sense of touch in the skin and play a role in transmitting sensory information to the brain.

Due to its rarity and potentially aggressive nature, individuals who suspect they may have a skin lesion that could be Merkel cell carcinoma should seek prompt medical

attention. Regular skin examinations and sun protection measures can also help reduce the risk of developing this type of skin cancer.

Clinical studies that explicitly target Merkel cell carcinoma are critical in determining the safety and efficacy of novel therapies for this illness. These studies are critical in establishing if novel medicines outperform established choices and provide substantial evidence to support their wider use.

This study focuses on the experiences of persons diagnosed with Merkel cell carcinoma while they actively participate in a unique clinical trial involving medicinal therapies. The major focus is on closely monitoring trial completion rates and voluntary withdrawals among these individuals.

## Exploring the Essence of Observational Studies

Participating in this medical trial immerses you in an observational study, a subset of clinical research that is precisely designed to gain insights via the undisturbed monitoring of patients while maintaining their care plans.

Researchers will only observe your trip, methodically examining the consequences of your condition without making any changes. This particular trial design is critical in improving our understanding of the intrinsic evolution of a given medical illness and its influence on persons who have it. By actively participating in this observational study, you greatly help to broaden the boundaries of medical knowledge and stimulate improvements in the care offered to patients suffering from the same ailment.

# Comparing This Trial to Other Merkel Cell Carcinoma Clinical Studies

It is critical to recognize the uniqueness of this clinical experiment. It operates on an observational basis, which means that your participation will not include the delivery of particular therapies or interventions. Understanding the complete spectrum of Merkel cell carcinoma clinical trials, including interventional studies in which participants follow particular treatment procedures, is critical.

Making an educated decision regarding possible clinical trial participation demands an active strategy that includes researching and evaluating various trials. Clinicaltrials.gov and other platforms provide a plethora of information about <u>research relevant to Merkel</u> cell carcinoma. Furthermore, Power's specialized web platform provides a complete

listing of ongoing <u>Merkel cell carcinoma clinical trials</u> that are actively recruiting volunteers. You empower yourself to confidently design your participation decision by completing comprehensive research and developing a profound awareness of various clinical trial models.

## **Engaging Actively in Clinical Trial Surveys**

We cordially invite you to actively share your experiences within the context of this observational clinical investigation. This initiative requires you to complete surveys every two weeks, which will take roughly 20-30 minutes of your valuable time. Furthermore, we stand ready to conduct check-in calls at quarterly intervals, a commitment that will last the life of your participation in the trial.

It is critical to emphasize that your participation in the survey portion of the study is completely optional. You have the freedom to choose whether to answer select questions or the complete questionnaire. Furthermore, you have the freedom to discontinue your participation in the trial whenever you choose. Recognizing that the choice to enroll in a clinical study is extremely personal, we are committed to providing the appropriate assistance. Your privacy and comfort remain our top considerations, and we are committed to respecting and supporting your decision-making process throughout the trial.

# Ensuring the Confidentiality of Your Responses

Maintaining the strictest confidentiality of your information is critical during the duration of this research investigation. We kindly request that you refrain from entering any personal or identifiable information in your questionnaire replies to protect your anonymity. The committed research team is unwavering in their dedication to enhancing the safety of your anonymity. Nonetheless, it is critical to recognize that special legal circumstances may emerge that require the disclosure of personal data.

#### Potential Risks

While clinical trials contribute greatly to medical advancement, it is critical to recognize the possible health concerns that participants may suffer, especially in studies investigating innovative medicines.

Our observational clinical research, on the other hand, takes a different strategy, proactively reducing these risks by not providing new therapies to participants. Instead, we place a premium on rigorous monitoring and result evaluation to eliminate avoidable health risks.

#### **Envisioned Benefits**

Though the immediate advantages for those participating in this observational clinical research may not be obvious, their participation has the potential to affect others. The data collected from participants will be used to improve future approaches for recruiting people with Merkel cell carcinoma, potentially widening the scope of medical study. Individuals who start on this clinical journey might act as catalysts for revolutionary change in the domain of medical research, perhaps changing the path for future Merkel cell carcinoma sufferers.

### Navigating the Depths of Diversity in Clinical Trials

For individuals with a keen interest in unraveling the complicated tapestry of representation inside clinical trials, a variety of internet resources awaits your active participation.

Whether your objective is to comprehend the intricacies of obstacles and opportunities surrounding clinical trial inclusion, or you just want to broaden your personal knowledge, the following resources might be helpful:

Westen, Drew I., Shannon Wiltsey Stirman, and Robert J. DeRubeis. "Are research patients and clinical trials representative of clinical practice?." (2006).

Tao, Cui, Guoqian Jiang, Weiqi Wei, Harold R. Solbrig, and Christopher G. Chute.

"Towards semantic-web based representation and harmonization of standard meta-data models for clinical studies." *AMIA summits on translational science proceedings* 2011 (2011): 59.

#### Confirmation of Informed Consent

I hereby certify that I have spent substantial time studying and internalizing the information included in the informed consent form, either via self-guided exploration or with the assistance of a trusted individual who has expressed its essence to me. All of my concerns and anxieties have been thoroughly handled to my complete satisfaction.

I am well aware that my participation in this study is the consequence of my own free will, and I retain the only right to withdraw my permission without rationale or financial repercussions. It has been made clear to me that a duplicate of this informed consent form will be provided for my own records.

After careful consideration and evaluation of the material supplied to me, I hereby give my permission to participate in this study, indicating my informed and autonomous decision.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

## Confirmation from Informed Consent Facilitator

I now confirm unequivocally that I participated in a long discourse with the participant, gradually revealing the complexities contained within this written paper. My major goal was to ensure that the patient understood the research's broad aims, methodology used, potential risks and benefits, and other critical components inherent to the Merkel cell carcinoma clinical trial.

Ample room was made available for the participant, which encouraged the development of questions and facilitated the explanation of ambiguities or misconceptions. It is critical to underline that his or her participation in this trial is the result of their voluntary decision, and they have the ultimate right to withdraw at any time, for any reason, without incurring any financial responsibilities.

Following the participant's grant of consent, they were given a scrupulously kept replica of this written document, which acted as a repository for their particular records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| <br>Date |